CLINICAL TRIAL: NCT06484816
Title: A Dose Escalation and Expansion Phase I Study Evaluating the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of TGRX-1942 in Patients with Advanced Solid Tumor And/or Relapsed/Refractory Hematologic Malignancies
Brief Title: TGRX-1942 Chinese Phase I for Advanced Solid Tumor And/or Relapsed/Refractory Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen TargetRx, Inc. (Industry)
Collaborators: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGRX-1942-1001
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Non Small Cell Lung Cancer; Advanced Solid Tumor; Hematologic Malignancy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: TGRX-1942 (Experimental): Patients will be given one of the doses of 4mg, 10mg, 20mg, 30mg, 40mg, 50mg, or 60mg orally once a day
  Interventions: Drug: TGRX-1942

INTERVENTIONS:
Drug: TGRX-1942 — At dose escalation phase, TGRX-1942 will be given orally to patient once a day under a 7-dose sequence of 4mg, 10mg, 20mg, 30mg, 40mg, 50mg, and 60mg. The dose level a particular patient will be assigned depends on the progression of the study and PI evaluation on the safety of previous dose group(s).

SUMMARY:
A phase I study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of TGRX-1942 in patients with advanced solid tumor and/or relapsed or refractory hematological malignancies

DETAILED DESCRIPTION:
This study is designed as a three-part study, with dose escalation, dose expansion and indication expansion phases. Patients with advanced solid tumors will be initially enrolled to the study. Other indications including solid tumors with specific gene mutations, or other hematological malignancies with be considered for expansion phases, with appropriate doses as evaluated at the end of dose escalation phase.

ELIGIBILITY:
Inclusion Criteria:

* For dose escalation phase, patient is diagnosed with advanced/metastatic solid tumor who had failed standard therapies and does not have available effective treatment, or who relapsed from prior treatments
* ECOG score of equals to or lower than 1
* Life expectancy of at least 3 months
* Adequate systemic and organ functions, including hematologic, hepatic and kidney functions
* Willing to provide available tumor biopsy sample or reports, or willing to undergo tumor biopsy examination, and willing to partake whole blood sampling for evaluations
* For female of child-bearing potential, willing to undergo plasma pregnancy test 28 days before first dose and have negative results
* Male and Female of child-bearing potential must agree to take effective contraceptive measures during the entire treatment period and for 2 months after the end of treatment
* Understand and willing to sign informed concent; willing and able to complete the visiting schedule and other tasks as required for the study

Exclusion Criteria:

* Allergic to any of the ingredient of the investigational drug
* History of other primary malignancies
* Have adverse/toxic effects from previous treatment that has not recovered to CTCAE 5.0 <= Grade 1
* Received other anti-tumor treatments (i.e., chemotherapy, biologics, immunotherapy, targeted therapy, etc.) 28 days before first dose, or radiation therapy 14 days before first dose
* Used drugs known to significantly affect P450 metabolism 2 weeks before first dose
* Participated in other clinical trials and used other investigational agents 28 days before first dose
* Received major surgeries or had traumatic injuries 28 days before first dose
* Need to use concomitant drugs that could cause QTc elongation or induce Torsades de Pointes
* History or presence of other medical conditions, such as HIV/HBV/HCV positive; received anticoagulation treatment; coagulation dysfunction; major or clinically significant cardiovascular disease; pneumonia; clinically significant gastrointestinal abnormalities that could affect drug absorption; uncontrollable hypertension; ulcer in abdomen, intestine, stomach, trachea or esophagus; uncontrolled seizure or have other central nervous system diseases, poorly managed diabetes; long QT syndrome; uncontrolled active infections; uncontrolled pericardial or abdominal effusion; adrenaline malfunction; thyroid dysfunction; severe unhealed wound, ulcer or bone fractures; Toxic epidermal necrolysis; Stevens-Johnson syndrome
* Have symptomatic or uncontrolled primary or metastatic central nervous system tumor or Leptomeninges tumor, or untreated diseases that cause compressions to spinal cords
* For female patients: in pregnancy or breast-feeding periods
* Presence of any condition or history that could affect study results or participation to the study in the judgement of the investigator
* Used immunosuppressant drugs within14 days before first dose
* Received vaccine injection within 30 days of Cycle 1 Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events/serious adverse events | From screening through completion of the study, an average of 3.5 years.
  to record and analyse the occasions and rates of subjects with adverse events (AEs) and serious adverse events (SAEs) to understand drug safety profile
Maximum Tolerated Dose (MTD) | From Day 1 of Cycle 1 to Day 28 of Cycle 1 of dose escalation phase (each cycle is 28 days)
  MTD is defined as the dose level with dose-limiting toxicity (DLT) rate of greater than 0.322 as calculated using the BOIN design at dose escalation phase.

SECONDARY OUTCOMES:
Preliminary efficacy | From screening, every 3 cycles during treatment period (each cycle is 28 days) and at end of study, an average of 3.5 years.
  For patients with advanced solid tumors, efficacy is evaluated based on RECIST 1.1 criteria which evaluates tumor size changes. Preliminary efficacy is evaluated by Principal investigator.
Time to Maximum Concentration (Tmax) | On day 1-6 of the single dosing phase; patient will only be dosed once on Day 1 of this phase
  To measure the time to reach maximum plasma drug concentration from dosing
Maximum Concentration (Cmax) | On day 1-6 of the single dosing phase; patient will only be dosed once on Day 1 of this phase
  To measure the maximum plasma drug concentration from dosing
Area Under Curve (AUC0-t) | On day 1-6 of the single dosing phase; patient will only be dosed once on Day 1 of this phase
  To calculate area under curve of drug plasma concentration from dosing to last measurable time point
Half life (T1/2) | On day 1-6 of the single dosing phase; patient will only be dosed once on Day 1 of this phase
  to measure the time needed to reach half maximal concentration from dosing
Apparent Clearance (CL/F) | On day 1-6 of the single dosing phase; patient will only be dosed once on Day 1 of this phase
  To calculate the rate of clearance of the drug after first dosing
Apparent Volume of Distribution (Vz/F) | On day 1-6 of the single dosing phase; patient will only be dosed once on Day 1 of this phase
  To calculate the volume of distribution of the drug after first dosing
Steady State Time to Maximal Concentration (Tmax,ss) | On day 1 of Cycle 1 of dose escalation phase (each cycle is 28 days)
  Under once daily dosing schedule, to measure the time to reach maximum plasma drug concentration between two dosing timepoints
Steady State Maximal Concentration (Cmax,ss) | On Day 1, 8, 15 and 22 of Cycle 1 and Day 1 of every 3 cycles (each cycle is 28 days). Average duration of the treatment period is 3 years.
  Under once daily dosing schedule, to measure the maximal plasma drug concentration from first dosing
Steady State Trough Concentration (Ctrough,ss) | On Day 1, 8, 15 and 22 of Cycle 1 and Day 1 of every 3 cycles (each cycle is 28 days). Average duration of the treatment period is 3 years.
  Under once daily dosing schedule, to measure the minimal plasma drug concentration from first dosing
Steady State Area Under Curve (AUC0-t,ss) | On Day 1, 8, 15 and 22 of Cycle 1 and Day 1 of every 3 cycles (each cycle is 28 days). Average duration of the treatment period is 3 years.
  Under once daily dosing schedule, to calculate area under curve of drug plasma concentration between two dosing timepoints

CONTACTS AND LOCATIONS:
Overall Officials: panhongming@zju.edu.cn Pan, MD, Principal Investigator — Zhejiang University School of Medicine Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China